CLINICAL TRIAL: NCT00627965
Title: Randomized, Controlled Trial of Regular Sildenafil Citrate in the Prevention of Altitude Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altitude Physiology Expeditions (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Director, Altitude Physiology Expeditions
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sildenafil1
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-02

CONDITIONS: High Altitude Pulmonary Edema; Acute Mountain Sickness
Keywords: Sildenafil citrate; Prevention; High Altitude Pulmonary Edema; Acute Mountain Sickness; Healthy Lowland Subjects; Pulmonary Artery Systolic Pressure
MeSH Terms: conditions — Altitude Sickness | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sildenafil citrate
  Interventions: Drug: Sildenafil citrate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil citrate — 50mg tds
  Arms: 1
Drug: Placebo — Placebo tds
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether regular oral use of sildenafil citrate can prevent or attenuate high altitude illnesses.

DETAILED DESCRIPTION:
High altitude pulmonary oedema (HAPE) is a life-threatening non-cardiogenic lung injury precipitated by exaggerated pulmonary hypertension. The incidence of this rapidly progressive illness, among the estimated 40 million visitors to high altitude each year, may be as high as 0.5-2.0%. The pathogenesis of HAPE is multifactorial and may include impaired clearance of alveolar fluid, increased pulmonary vascular permeability and genetic susceptibility. Elevated pulmonary artery pressure (PAP) caused by hypoxic pulmonary vasoconstriction (HPV) is a key prerequisite for the development of HAPE and thus the reduction of PAP is paramount in the prophylaxis and treatment of this devastating illness.

Nitric oxide (NO) is thought to play an important role in the exaggerated HPV that characterises HAPE. NO, constitutively produced in the lung by the enzyme endothelial nitric oxide synthase (eNOS), increases intracellular cGMP in pulmonary vascular smooth muscle and activates cGMP-dependent protein kinase, ultimately leading to a reduction in intracellular calcium and smooth muscle relaxation. HAPE-susceptible individuals exhale less NO during both normobaric and hypobaric hypoxia suggesting that a deficiency of NO synthesis may predispose to HAPE. At high altitude, inhaled NO causes a significantly greater reduction in the systolic PAP of HAPE-susceptible individuals compared to its effect on the PAP of HAPE-resistant subjects, but the administration of NO would be impractical in the field. Most recently, work has concentrated on another target in the NO pathway.

Sildenafil citrate is an orally active, potent and selective phosphodiesterase type-5 (PDE-5) inhibitor. PDE-5 is the predominant enzyme responsible for degradation of cGMP in the lung. In a small sea level study, Zhao et al. demonstrated that pre-treatment with sildenafil nearly completely abolished the pulmonary vasopressor response to breathing hypoxic gas in healthy humans. More recently, studies at altitude have also shown reductions in pulmonary artery systolic pressure (PASP) in subjects taking sildenafil at high altitude.

One potential problem with the use of sildenafil at altitude is that PDE-5 inhibitors may worsen symptoms of acute mountain sickness (AMS). Headache is a defining symptom in AMS and is a prominent side effect of sildenafil.

We conducted a double-blind placebo-controlled randomised trial to assess the effect of regular sildenafil administration on PASP and Lake Louise AMS score at an altitude of 5200 m.

ELIGIBILITY:
Inclusion Criteria:

* Participant in Apex 2 high altitude expedition

Exclusion Criteria:

* Previous history of high altitude pulmonary edema

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-03; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary Artery Systolic Pressure (PASP)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bates, Principal Investigator — Altitude Physiology Expeditions

REFERENCES:
- [Derived] MacCormick IJ, Somner J, Morris DS, MacGillivray TJ, Bourne RR, Huang SS, MacCormick A, Aspinall PA, Baillie JK, Thompson AA, Dhillon B. Retinal vessel tortuosity in response to hypobaric hypoxia. High Alt Med Biol. 2012 Dec;13(4):263-8. doi: 10.1089/ham.2011.1097. PMID 23270443
- [Derived] Bates MG, Thompson AA, Baillie JK, Sutherland AI, Irving JB, Hirani N, Webb DJ. Sildenafil citrate for the prevention of high altitude hypoxic pulmonary hypertension: double blind, randomized, placebo-controlled trial. High Alt Med Biol. 2011 Fall;12(3):207-14. doi: 10.1089/ham.2011.0007. PMID 21962063
- See also: Research group website coordinating future studies — http://altitude.org